CLINICAL TRIAL: NCT03161600
Title: Improving Surgical/Medical Oncology Collaboration for Breast Cancer Treatment Planning: Pilot Testing the Impact of Continuing Education and Patient Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: G402
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Carevive CPS — This intervention will focus on the use of the Carevive CPS at a surgical visit, enabling providers to deliver evidence-based and personalized treatment care plans to their breast cancer patients. The Carevive CPS collects electronic patient reported outcomes (ePROS) and clinical data, reported and generated by clinical staff and/or extracted from the electronic medical record (EMR), and uses these to auto-generate the personalized care plans. Care plan content is drive by practice guidelines and other peer-reviewed evidence, and includes patient education, resources, and referrals developed by cancer clinicians and researchers.

SUMMARY:
This study will explore provider's screening and management practices for eligibility for neoadjuvant therapy from baseline to following the project intervention (use of a novel existing technology, the Carevive Care Planning System at the point of care plus provider continuing medical education.

DETAILED DESCRIPTION:
The overarching goals are to improve clinician knowledge about evidence-based practices for neoadjuvant therapy for breast cancer, increase appropriate referrals to medical oncology for consideration of preoperative systemic therapy (as determined by adherence to NCCN pre-operative systemic therapy guidelines), and to improve communication between the multidisciplinary team and patient regarding the appropriateness, selection, and timing of neoadjuvant therapy. Secondary objectives include a) evaluation of the impact of the intervention on actual prescription of neoadjuvant therapy to eligible patients and b) evaluation of the impact of the intervention on surgeons and medical oncologists' knowledge, attitudes, and beliefs about the benefits of neoadjuvant therapy. We will also explore the acceptability and utilization of the Carevive care plan during medical oncologists' initial consultations after referral of patients from surgical practices. In this project, 25 newly diagnosed breast cancer patients will be recruited over a 3-6 month period, screened for eligibility for neoadjuvant therapy, and assessed for patient treatment preferences at time of surgical consultation using a novel and commercially available electronic technology, the Carevive Care Planning System (CPS). Patients will receive a care plan that explains neoadjuvant therapy among possible treatment options. In addition, patients will be screened for distress as well as eligibility for genetic counseling (according to NCCN referral criteria) and fertility preservation (according to ASCO guidelines) referrals, and the Carevive care plans provided will also incorporate personalized referrals to these related services where applicable.

Retrospective chart reviews (from both surgical and medical oncology practices participating in this project), complemented by data extracted from the Carevive CPS, will be used to assess changes in rates of referrals to medical oncology for discussion and actual prescriptions of neoadjuvant therapy, as compared to historical data from prior publications documenting low rates of referral to, and receipt of, neoadjuvant therapy. Provider questionnaires exploring knowledge, attitudes, and beliefs about the benefits of neoadjuvant therapy will be completed at baseline and again at follow-up (≤4 weeks following intervention visit of their last patient) and changes will be explored using a pre-/post-test design. Use of a care planning technology to provide tailored education and individualized information may provide an easy, accessible and effective way to improve provider abilities to proactively identify patients eligible for specific therapies, understand patient treatment goals, concerns, drive shared decision making (SDM) and sufficiently collaborate with the multi-disciplinary team to provide optimal care.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18 years of age and older
* 2) Patients must have a diagnosis of breast cancer for which they must not have received or been scheduled for primary breast surgery at time of project intervention, and must be eligible for surgical resection (i.e. Stage I-III).

Exclusion Criteria:

* Any patient who cannot understand written or spoken English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Rates of provider self-report and actual percent of eligible patients referred to medical oncology for discussion of neoadjuvant therapy. | Year 1
  Data collected via chart abstraction and provider surveys will be analyzed.
Rates of actual prescription of neoadjuvant therapy to eligible patients | Year 1
  Data will be collected via chart abstraction

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No